CLINICAL TRIAL: NCT04197531
Title: A Comparative Evaluation of the Effect of EndoActivator and Endodontic Syringe Usage on Postoperative Pain in Root Canal Irrigations in Primary Molar Teeth: A Randomized Clinical Study
Brief Title: Postoperative Pain After the Use of Different Last Irrigation Method During Root Canal Treatment in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Husniye Gumus, Study Director, PHD., Dr., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/152
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Post Operative Pain
Keywords: EndoActivator; Irrigation; Postoperative pain; Primary teeth
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoActivator (Experimental)
  Interventions: Other: Irrigation Method
- Conventional Endodontic Syringe (Experimental)
  Interventions: Other: Irrigation Method

INTERVENTIONS:
Other: Irrigation Method — Irrigation Method

SUMMARY:
This study was to evaluate and compare the postoperative pain levels after using EndoActivator and conventional endodontic syringe irrigation in root canal therapy of primary molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients exhibiting positive or definitely positive behavior on the Frankl's behavior rating scale (rating 3 or 4 on the Frankl's scale)
* American Society of Anesthesiologists class 1 patients aged 5-9 years
* Patients with symptomatic irreversible pulpitis of maxillary primary molars confirmed using periapical radiographs, percussion, and cold test
* Patients having teeth with two-thirds of each root remaining
* Absence of periapical lesions and interradicular radiolucency
* Moderate to very severe (2-4) five-face scale pain scores in the 24-hour period before the procedure.

Exclusion Criteria:

* Patients who had taken analgesics and antibiotics within the last 12 hours before root canal treatment
* Teeth with pathologic root resorption
* Teeth with excessive mobility.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Pain level comparison after root canal treatment with two different irrigation methods:The five-face pain scale chart at 8th hours | 8th hours
  Pain levels according to the five-face scale were recorded numerically as no pain (0), mild pain (1), moderate pain (2), severe pain (3), or very severe pain (4). All participants and their parents were informed by a blind researcher about filling out the five-face pain scale chart. To achieve standardization, pain levels were recorded by the participants under the same parent's guidance at each time interval.
Pain level comparison after root canal treatment with two different irrigation methods:The five-face pain scale chart at 24th hours | 24th hours
  Pain levels according to the five-face scale were recorded numerically as no pain (0), mild pain (1), moderate pain (2), severe pain (3), or very severe pain (4). All participants and their parents were informed by a blind researcher about filling out the five-face pain scale chart. To achieve standardization, pain levels were recorded by the participants under the same parent's guidance at each time interval.
Pain level comparison after root canal treatment with two different irrigation methods:The five-face pain scale chart at 48th hours | 48th hours
  Pain levels according to the five-face scale were recorded numerically as no pain (0), mild pain (1), moderate pain (2), severe pain (3), or very severe pain (4). All participants and their parents were informed by a blind researcher about filling out the five-face pain scale chart. To achieve standardization, pain levels were recorded by the participants under the same parent's guidance at each time interval.
Pain level comparison after root canal treatment with two different irrigation methods:The five-face pain scale chart at 72th hours | 72th hours
  Pain levels according to the five-face scale were recorded numerically as no pain (0), mild pain (1), moderate pain (2), severe pain (3), or very severe pain (4). All participants and their parents were informed by a blind researcher about filling out the five-face pain scale chart. To achieve standardization, pain levels were recorded by the participants under the same parent's guidance at each time interval.

SECONDARY OUTCOMES:
Analgesic intake comparison after root canal treatment with two different irrigation methods at 0-8 hours. | 0-8 hours
  The patients were asked to choose one of the two options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep".
Analgesic intake comparison after root canal treatment with two different irrigation methods at 8-24 hours. | 8-24 hours
  The patients were asked to choose one of the two options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep".
Analgesic intake comparison after root canal treatment with two different irrigation methods at 24-48 hours. | 24-48 hours
  The patients were asked to choose one of the two options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep".
Analgesic intake comparison after root canal treatment with two different irrigation methods at 48-72 hours. | 48-72 hours
  The patients were asked to choose one of the two options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep".

CONTACTS AND LOCATIONS:
Overall Officials: Hüsniye Gümüş, PHD., Dr., Study Director — Erciyes University, Faculty of Dentistry
Locations (1):
- Erciyes University, Faculty of Dentistry, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramamoorthi S, Nivedhitha MS, Divyanand MJ. Comparative evaluation of postoperative pain after using endodontic needle and EndoActivator during root canal irrigation: A randomised controlled trial. Aust Endod J. 2015 Aug;41(2):78-87. doi: 10.1111/aej.12076. Epub 2014 Sep 4. PMID 25195661
- [Background] Yilmaz K, Tufenkci P, Adiguzel M. The effects of QMix and EndoActivator on postoperative pain in mandibular molars with nonvital pulps: a randomized clinical trial. Clin Oral Investig. 2019 Nov;23(11):4173-4180. doi: 10.1007/s00784-019-02856-6. Epub 2019 Feb 27. PMID 30815731
- [Derived] Gumus H, Delikan E. The effect of sonic activation of irrigant on postoperative pain after root canal treatment in primary molar teeth: a randomized, clinical study. Clin Oral Investig. 2021 Jan;25(1):363-370. doi: 10.1007/s00784-020-03687-6. Epub 2020 Nov 12. PMID 33184717